CLINICAL TRIAL: NCT05833100
Title: Method Comparison/User Evaluation of the i-SENS Self-Monitoring Blood Glucose / β-Ketone System (CareSens PRO GK BT)
Brief Title: Method Comparison/User Evaluation of the i-SENS Self-Monitoring Blood Glucose / β-Ketone System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a change in the marketing strategy of the device.
Sponsor: i-SENS, Inc. (Industry)
Collaborators: Avania (Industry); Rainier Clinical Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BGM-2205084
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-01

CONDITIONS: Diabetes
Keywords: Self-Monitoring Blood Glucose (SMBG)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: A minimum of 350 different subjects, both naive and non-naive SMBG users, is required. At least 10% of the study participants should be naive to SMBGs and may include non-diabetic subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Users of the Blood Glucose/b-Ketone Monitoring System (Experimental): Participants are individuals who have either been diagnosed with diabetes or not and are naive users of CareSens PRO GK BT.
  Interventions: Device: CareSens PRO GK Blood Glucose/b-Ketone Monitoring system

INTERVENTIONS:
Device: CareSens PRO GK Blood Glucose/b-Ketone Monitoring system — All BG results were compared to YSI 2300 reference method results obtained from subjects' capillary blood.
  All Ketone results were compared to Randox Imola D-3-Hydroxybutyrate analyzer.

SUMMARY:
The goal of this clinical trial is to assess the accuracy and usability of the blood glucose meter in untrained participants, both with or without diabetes, as well as those with pre-diabetes.

DETAILED DESCRIPTION:
Participants will personally date and sign the informed consent before engaging in any study-related activity. Participants use a single-use lancing device to lance their finger and perform a blood glucose test with glucose test strips on the meter. Trained staff collects more blood samples for YSI and hematocrit measurement (approx. 300-350μL) using a specified lancet within 5 minutes of the first evaluable meter reading. Follow the same process to measure Ketones using the β-Ketone test strip on the same meter. The staff collects more blood samples for Imola and hematocrit measurement (approx. 500-550μL).

After subjects have completed the testing, they are then asked to complete usability questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and older
* People with type 1 diabetes, type 2 diabetes, pre-diabetes and no diabetes (self- reported)
* Able to speak, read and understand English (subjects must demonstrate ability to read a sentence from a page of the draft device labeling instructions (user's manual) to qualify for the study)
* Willing to complete all study procedures
* Has read, understood, and signed the Informed Consent Form

Note: The study group consists of naive SMBG users and non-naive SMBG users. At least 10% of study participants should be naive for SMBG, including subjects without diabetes.

Exclusion Criteria:

* Hemophilia or any other bleeding disorder
* Works for a medical laboratory, hospital, other clinical setting or a medical device company that involves training on or clinical use of blood glucose meters
* Physical, visual or neurological impairments as determined by the investigator or designee that would make the subject unable to perform self-testing (reason for exclusion will be clearly documented by investigator or designee directly on the subject disposition form)
* A condition, which in the opinion of the investigator or designee, would put the subject or study conduct at risk (reason for exclusion will be clearly documented by investigator or designee on the subject disposition form).

Note 1: In the event of a physical, visual or neurological impairment that makes it difficult for a subject to complete the questionnaire, the subject's verbal responses will be accepted and should be appropriately documented as such within the subject records form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rainier Clinical Research Center, Renton, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 5 and 10 participants are enrolled per day at one site. A total of 76 participants were recruited in 11 sessions; 2 screening failed and 74 completed.
Pre-assignment Details: Termination resulted from a change in the marketing strategy of the clinical trial.
Groups:
- Users of the Blood Glucose Monitoring System (Only): Participants are individuals who have either been diagnosed with diabetes or not and are naive users of CareSens PRO GK BT.
  All BG results were compared to YSI 2300 reference method results obtained from subjects' capillary blood.
- Users of the Blood Glucose and b-Ketone Monitoring System: Participants are individuals who have either been diagnosed with diabetes or not and are naive users of CareSens PRO GK BT.
  All BG results were compared to YSI 2300 reference method results obtained from subjects' capillary blood. All Ketone results were compared to the Randox Imola D-3-Hydroxybutyrate analyzer.
- Users of the b-Ketone Monitoring System (Only): Participants are individuals who have either been diagnosed with diabetes or not and are naive users of CareSens PRO GK BT.
  All Ketone results were compared to Randox Imola D-3-Hydroxybutyrate analyzer.
Period: Day 1(August 15th)
Arm/Group | Users of the Blood Glucose Monitoring System (Only) | Users of the Blood Glucose and b-Ketone Monitoring System | Users of the b-Ketone Monitoring System (Only)
Started | 2 | 3 | 0
Completed | 2 | 3 | 0
Not Completed | 0 | 0 | 0
Period: Day 2(August 16th)
Arm/Group | Users of the Blood Glucose Monitoring System (Only) | Users of the Blood Glucose and b-Ketone Monitoring System | Users of the b-Ketone Monitoring System (Only)
Started | 5 | 0 | 0
Completed | 4 (This measurement was made in the con-sol mode. This data is excluded from analysis.) | 0 | 0
Not Completed | 1 | 0 | 0
Period: Day 3(August 23rd)
Arm/Group | Users of the Blood Glucose Monitoring System (Only) | Users of the Blood Glucose and b-Ketone Monitoring System | Users of the b-Ketone Monitoring System (Only)
Started | 5 | 3 | 0
Completed | 5 | 3 | 0
Not Completed | 0 | 0 | 0
Period: Day 4(August 24th)
Arm/Group | Users of the Blood Glucose Monitoring System (Only) | Users of the Blood Glucose and b-Ketone Monitoring System | Users of the b-Ketone Monitoring System (Only)
Started | 0 | 2 | 0
Completed | 0 | 2 | 0
Not Completed | 0 | 0 | 0
Period: Day 5(August 29th)
Arm/Group | Users of the Blood Glucose Monitoring System (Only) | Users of the Blood Glucose and b-Ketone Monitoring System | Users of the b-Ketone Monitoring System (Only)
Started | 0 | 5 | 1
Completed | 0 | 5 | 1
Not Completed | 0 | 0 | 0
Period: Day 6(August 31st)
Arm/Group | Users of the Blood Glucose Monitoring System (Only) | Users of the Blood Glucose and b-Ketone Monitoring System | Users of the b-Ketone Monitoring System (Only)
Started | 0 | 6 | 0
Completed | 0 | 6 | 0
Not Completed | 0 | 0 | 0
Period: Day 7(September 6th)
Arm/Group | Users of the Blood Glucose Monitoring System (Only) | Users of the Blood Glucose and b-Ketone Monitoring System | Users of the b-Ketone Monitoring System (Only)
Started | 0 | 7 | 1
Completed | 0 | 7 | 1
Not Completed | 0 | 0 | 0
Period: Day 8(September 9th)
Arm/Group | Users of the Blood Glucose Monitoring System (Only) | Users of the Blood Glucose and b-Ketone Monitoring System | Users of the b-Ketone Monitoring System (Only)
Started | 0 | 8 | 0
Completed | 0 | 8 | 0
Not Completed | 0 | 0 | 0
Period: Day 9(September 13th)
Arm/Group | Users of the Blood Glucose Monitoring System (Only) | Users of the Blood Glucose and b-Ketone Monitoring System | Users of the b-Ketone Monitoring System (Only)
Started | 0 | 10 | 0
Completed | 0 | 10 | 0
Not Completed | 0 | 0 | 0
Period: Day 10(September 19th)
Arm/Group | Users of the Blood Glucose Monitoring System (Only) | Users of the Blood Glucose and b-Ketone Monitoring System | Users of the b-Ketone Monitoring System (Only)
Started | 0 | 8 | 0
Completed | 0 | 8 | 0
Not Completed | 0 | 0 | 0
Period: Day 11(September 21st)
Arm/Group | Users of the Blood Glucose Monitoring System (Only) | Users of the Blood Glucose and b-Ketone Monitoring System | Users of the b-Ketone Monitoring System (Only)
Started | 0 | 8 | 0
Completed | 0 | 8 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The order of measurements is as follows: PRO GK (BG) > YSI > PRO GK (b-Ketone) > Randox
  For BG monitoring system analysis excluding
  * Console mode measurements (#8)
  * CRF not confirmed & staff unable to collect 300uL blood (#23)
  * YSI calibration fail (#41)
  For b-Ketone monitoring system analysis excluding
  * Measurement with glucose strips (#7)
  * Console mode measurements (#8)
  * Randox value <0.07 (#2,5,6,9,10,12,13,15,17,18)
Groups:
- Users of the Blood Glucose Monitoring System (Only): Untrained subjects used the CareSens Pro GK Blood Glucose/b-Ketone Monitoring System.
  All BG results were compared to YSI 2300 reference method results obtained from subjects' capillary blood.
- CareSens Pro GK Blood Glucose and b-Ketone Monitoring System.: Untrained subjects used the CareSens Pro GK Blood Glucose/b-Ketone Monitoring System.
  BG and b-Ketone results from PRO GK were compared to YSI 2300 and the Randox Imola D-3-Hydroxybutyrate analyzer.
- Users of the b-Ketone Monitoring System (Only): Untrained subjects used the CareSens Pro GK Blood Glucose/b-Ketone Monitoring System.
  All Ketone results were compared to the Randox Imola D-3-Hydroxybutyrate analyzer.
- Total: Total of all reporting groups
Arm/Group | Users of the Blood Glucose Monitoring System (Only) | CareSens Pro GK Blood Glucose and b-Ketone Monitoring System. | Users of the b-Ketone Monitoring System (Only) | Total
Number analyzed (Participants) | 11 | 60 | 2 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 33 | 0 | 43
  >=65 years | 1 | 27 | 2 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 39 | 1 | 45
  Male | 6 | 21 | 1 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 58 | 0 | 60
  Not Hispanic or Latino | 9 | 2 | 2 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 8 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 1 | 7 | 0 | 8
  White | 8 | 42 | 2 | 52
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Conditions [Number; unit: participants]
  Type 1 Diabetes | 4 | 20 | 0 | 24
  Type 2 Diabetes | 6 | 37 | 2 | 45
  Pre-Diabetes | 0 | 0 | 0 | 0
  No Diabetes | 1 | 3 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Hematocrit Measurement
Description: The subject's hematocrit measurement should be within the range of 20-60% for the result to be considered evaluable. Two consecutive measurements are taken, and it determinds the analytical validity of a blood sample by the average value.
Time Frame: The blood sample is immediately collected for hematocrit measurement within 5 minutes of the first evaluable BG meter reading and then, centrifuge the sample within 10 minutes of sample collection.
Population: BG monitoring system data excludings>
  * Console mode measurements (#8)
  * CRF has not been confirmed & staff is unable to collect 300uL of blood sample (#23)
  * Screening fail (#30,33)
  * YSI calibration fail (#41)
    b-Ketone monitoring system data excludings>
  * Randox value <0.07 for weeks 1 and 2 (#2,5,6,9,10,12,13,15,17,18)
  * Measurement with glucose strips (#7)
  * Console mode measurements (#8)
  * Screening fail (#30,33)
Measure: Mean (Full Range); unit: Percentage of hematocrit
Groups:
- Users of the Blood Glucose Monitoring System: Untrained subjects with diabetes used the CareSens Pro GK Blood Glucose/b-Ketone Monitoring System.
  CareSens PRO GK Blood Glucose/b-Ketone Monitoring system: All BG results were compared to YSI 2300 reference method results obtained from subjects' capillary blood.
- Users of the b-Ketone Monitoring System: Untrained subjects with diabetes used the CareSens Pro GK Blood Glucose/b-Ketone Monitoring System.
  CareSens PRO GK Blood Glucose/b-Ketone Monitoring system: All Ketone results were compared to Randox Imola D-3-Hydroxybutyrate analyzer.
Arm/Group | Users of the Blood Glucose Monitoring System | Users of the b-Ketone Monitoring System
Number analyzed (Participants) | 71 | 62
Percentage of hematocrit
  1st meaasurement | 44.27 [36 to 52] | 44.10 [36 to 52]
  2nd measurement | 44.65 [36 to 53] | 44.65 [36 to 53]
  Average of duplicated measurements | 44.46 [36 to 52.5] | 44.56 [36 to 52.5]

2. Secondary Outcome: Glucose Testing of Subject Plasma Samples
Description: The subject capillary plasma samples will be tested in duplicate. If the average of replicates 1&2 do not fall within range (within 4% for readingsabove100mg/dL or 4 mg/dL for samples less than or equal to 100mg/dL) the sample will be run a third time and the 2 average replicate readings that fall within range (4% for readings above 100mg/dL or 4 mg/dL for samples less than or equal to 100mg/dL) will be recorded as evaluable.
  In general, duplicates will be averaged for each subject. If the sample is insufficient or missing and have only a single YSI value, it will be used as the YSI determination. If none of the 3 average replicates fall within (4% for readings above 100mg/dL or 4 mg/dL for samples less than or equal to 100mg/dL) will be recorded as non-evaluable. If the YSI autocals between subject sample duplicates, then another YSI 2747 standard will be run before completing the subject sample cycle.
Time Frame: Within 20 minuates of centrifugation
Reporting Status: Not Posted

3. Secondary Outcome: β-Ketone Testing of Subject Plasma Samples
Description: The subject capillary plasma sample will be tested in duplicate using Rx Imola analyzer. If the measured values differ by > 0.075 mmol/L at ketone < 1.5 mmol/L or > 5% at ketone ≥ 1.5 mmol/L, the sample will be run a third time and the 2 average replicate readings that fall within range will be recorded as evaluable. In general, duplicates will be averaged for each subject. If the sample is insufficient or missing and has only a single Rx Imola value, it will be used as the Rx Imola determination. If none of the 3 average replicates fall within > 0.075 mmol/L at ketone < 1.5 mmol/L or > 5% at ketone ≥ 1.5 mmol/L for readings, it will be recorded as non-evaluable.
Time Frame: Within 20 minuates of centrifugation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Users of the Blood Glucose Monitoring System: Participants are individuals who have either been diagnosed with diabetes or not and are naive users of CareSens PRO GK BT.
  All BG results were compared to YSI 2300 reference method results obtained from subjects' capillary blood.
- Users of the Blood b-Ketone Monitoring System: Participants are individuals who have either been diagnosed with diabetes or not and are naive users of CareSens PRO GK BT.
  All Ketone results were compared to Randox Imola D-3-Hydroxybutyrate analyzer.
Arm/Group | Users of the Blood Glucose Monitoring System | Users of the Blood b-Ketone Monitoring System
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/62
Other Adverse Events (participants affected / at risk) | 0/71 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT05833100/Prot_SAP_002.pdf
  • Informed Consent Form (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT05833100/ICF_001.pdf